CLINICAL TRIAL: NCT04983121
Title: Efficacy and Safety of Pyrotinib Maleate Combined With ARX788 Neoadjuvant Treatment in Stage II-III HER2-positive Breast Cancer Patients Who Have Poor Outcomes After Treatment With Trastuzumab and Pertuzumab
Brief Title: Efficacy and Safety of Pyrotinib Maleate Combined With ARX788 Neoadjuvant Treatment in Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Director, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shengjing-LCG009
Record Dates: First submitted 2021-07-09; First posted 2021-07-30 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; Pyrotinib; Neoadjuvant treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — ARX788

STUDY DESIGN:
Intervention Model Description: Single Group: single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combine treatment group (Experimental): This study adopts a single-arm, multi-center, open design. As per the initial plan, 30 stage II-III human epidermal growth factor receptor 2(HER2)-positive breast cancer patients who have received neoadjuvant therapy containing trastuzumab and pertuzumab and have been assessed as stable disease (SD) during the neoadjuvant treatment (an increase of 0-20%), disease progression (PD), inoperable or failing to meet the breast-conserving requirements will be enrolled to receive pyrotinib combined with Next-generation Site-specific HER2-targeting Antibody-drug Conjugate (ARX788) neoadjuvant therapy. The main purpose of the study is to observe the efficacy and safety of pyrotinib combined with ARX788 neoadjuvant treatment in stage II-III HER2-positive breast cancer.
  Interventions: Drug: Next-generation Site-specific human epidermal growth factor receptor 2 (HER2)-targeting Antibody-drug Conjugate (ARX788)

INTERVENTIONS:
Drug: Next-generation Site-specific human epidermal growth factor receptor 2 (HER2)-targeting Antibody-drug Conjugate (ARX788) — The subjects who sign an informed consent will enter the treatment period after screening. Each eligible subject will receive pyrotinib, 320 mg once a day, with 21 days as a session, for 6 sessions in total before operation. Next-generation Site-specific human epidermal growth factor receptor 2 (HER2)-targeting Antibody-drug Conjugate (ARX788) will be intravenously injected at a dose of 1.5 mg/kg, once every 3 weeks, with 21 days as a session, for 6 sessions before surgery. Breast MRI and other imaging examinations will be reviewed every 2 sessions to evaluate the curative effect, and the patient's baseline will be defined based on the imaging report at the time of enrollment. If a definite effect (complete response/partial response) is achieved, surgical treatment will be performed within 4 weeks (> 2 weeks) after completion of 6 sessions of neoadjuvant therapy.
  Other Names: pyrotinib maleate

SUMMARY:
Next-generation Site-specific human epidermal growth factor receptor 2 (HER2)-targeting Antibody-drug Conjugate (ARX788) is an antibody-conjugated drug. Results from the phase I safety, tolerability and pharmacokinetic trial of ARX788 single drug in Chinese patients with advanced HER2 breast cancer indicated a good safety of the test drug, and responses to anti-tumor therapy were observed in the target dose group. Phase II clinical trial is being carried out gradually. This trial is designed to observe the effectiveness and safety of pyrotinib maleate combined with ARX788 neoadjuvant treatment in stage II-III HER2-positive breast cancer patients experiencing a poor efficacy of trastuzumab and pertuzumab.

DETAILED DESCRIPTION:
This study adopts a single-arm, multi-center, open design. As per the initial plan, 30 stage II-III human epidermal growth factor receptor 2 (HER2)-positive breast cancer patients who have received neoadjuvant therapy containing trastuzumab and pertuzumab and have been assessed as stable disease (SD) during the neoadjuvant treatment (an increase of 0-20%), disease progression (PD), inoperable or failing to meet the breast-conserving requirements will be enrolled to receive pyrotinib combined with Next-generation Site-specific HER2-targeting Antibody-drug Conjugate (ARX788) neoadjuvant therapy. The main purpose of the study is to observe the efficacy and safety of pyrotinib combined with ARX788 neoadjuvant treatment in stage II-III HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 but ≤ 75 years (The maximal age of the subjects enrolled in the Phase 3 study of pyrotinib is 75 years old, and there is no safety data for the use of the drug in older people);
* Diagnosis of breast cancer meets the following criteria: Histologically confirmed invasive breast cancer; Tumor staging: Stage II-III patients who meet the 8th edition of AJCC Cancer Staging Manual; Patients who have undergone neoadjuvant therapy with trastuzumab and pertuzumab and have been assessed as SD (an increase of 0-20%), PD, inoperable or failing to meet the breast-conserving requirements; Failing to meet the breast-conserving requirements is defined as not meeting the following criteria: tumor size of T1 and T2 stage, proper breast volume, proper tumor-to-breast volume ratio, and able to maintain a good breast shape after surgery.
* HER2-positive breast cancer pathologically confirmed is defined as Immunohistochemical method (IHC3+) or FISH+;
* Eastern Cooperative Oncology Group (ECOG) level 0-1;
* The functional level of major organs must conform to the following requirements: Neutrophils (ANC) ≥ 1.5×109/L (with no use of growth factors within 14 days); Platelet count (PLT) ≥ 100×109/L (with no correct treatment within 7 days ); Hemoglobin (Hb) ≥ 90 g/L (with no correct treatment within 7 days ); Total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN; Urea nitrogen and creatinine ≤ 1.5×ULN and creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula); Cardiac color Doppler ultrasound: left ventricular ejection fraction (LVEF) ≥ 50%; 12-lead electrocardiogram: QT interval ≤ 480 ms;
* Able to receive needle biopsy;
* Patients who participate in the trial voluntarily, sign an informed consent, have good compliance and are willing to comply with the follow-up visit.

Exclusion Criteria:

* Patients who are concurrently receiving other anti-tumor therapy;
* Bilateral breast cancer, inflammatory breast cancer, or occult breast cancer;
* With a history of any malignancies other than breast cancer in the past 5 years, excluding cured cervical carcinoma in situ, non-melanoma skin cancer or other malignant tumors;
* Inability to swallow, chronic diarrhea and intestinal obstruction, and having many factors that affect drug administration and absorption;
* Cardiac insufficiency, including but not limited to congestive heart failure, transmural myocardial infarction, angina pectoris requiring medical treatment, clinically significant valvular disease and high-risk arrhythmia, or abnormal QTc in the ECG examination during the screening period (at rest, QTc > 450 ms in male or QTc > 470 ms in female after correction of ECG examination);
* Uncontrolled hypertension (at rest, systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg);
* Patients who are suffering severe or uncontrolled systemic diseases, such as unstable or uncompensable respiratory, heart, liver, or kidney diseases, as per the investigator's judgments;
* Female patients during pregnancy and lactation, or those who are fertile and positive for baseline pregnancy test or those of childbearing age who are unwilling to take effective contraceptive measures throughout the trial period;
* Serious concomitant diseases or other comorbid diseases that will endanger the safety of patients or interfere with the completion of the trial, including but not limited to severe hypertension, severe diabetes mellitus, and active infections that are out of control;
* Patients with known allergies to any active ingredients or excipients of ARX788, or with a history of protein drug allergy, a history of specific allergies (asthma, rheumatism, eczematous dermatitis), or a history of other severe allergic reactions, who are unsuitable for ARX788 treatment as per the investigator's judgments;
* With a history of interstitial pulmonary disease, drug-induced pulmonary interstitial disease, and radiation pneumonitis that require hormone therapy, or any clinically active pulmonary interstitial disease as suggested by any evidence;
* Patients who are currently suffering from keratitis, corneal disease, retinal disease, or active eye infection that require any interventions for the eyes.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Residual tumor burden (RCB) classification in grades | At least 3 years since enrollment
  Postoperative pathological results will be used to assess the residual tumor area of primary breast tumor (area in mm×mm), the cell density of the residual tumor（cell density in percentages）, the proportion of carcinoma in situ (proportion of carcinoma in percentages), the number of positive lymph nodes and the diameter of largest metastasis with residual nodes (diameter in mm). The RCB class can be estimated from the above five pathological parameters through a network calculation: RCB-0 in grades: pCR; RCB-I in grades: minimal residual tumor; RCB-II: moderate residual tumor; RCB-III in grades: extensive residual tumor.

SECONDARY OUTCOMES:
Best overall response rate (BORR) in percentage | At least 3 years since enrollment
  The proportion of patients who achieve remission at any point during the study.
Total pathological complete response rate (tpCR) in percentage | At least 3 years since enrollment
  The standard for removal of breast and lymph node tumors which means there are no infiltrating cancer cells at the primary breast and axillary lymph nodes, and only intraductal cancer is allowed on the breast.
Total breast pathological complete remission rate (bpCR) in percentage | At least 3 years since enrollment
  The standard for breast and lymph node tumor removal which means that there are only infiltrating cancer cells at the primary breast tumor site.
Disease-free survival (DFS) | At least 3 years since enrollment
  the time from the day of enrollment to the first occurrence of recurrent disease, including second primary malignancies in the non-breast area and breast ductal carcinoma in situ.
Overall survival (OS) | At least 3 years since enrollment
  the time from the random date to death due to any cause.

OTHER OUTCOMES:
Adverse events (AE) | at least 3 years since enrollment
  Adverse events (AE) will be assessed as per the NCI-CTC AE 5.0 standard.

CONTACTS AND LOCATIONS:
Overall Officials: Cai-Gang Liu, Principal Investigator — Department of Breast Surgery, Shengjing Hospital affiliated to China Medical University
Locations (1):
- Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No